CLINICAL TRIAL: NCT01449695
Title: Nurse- and Web Based Intervention to Improve Medication Adherence in High Risk Cardiovascular Patients.
Brief Title: Intervention to Improve Medication Adherence in Cardiovascular Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Bas Bredie, MD, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 34338
Record Dates: First submitted 2011-10-05; First posted 2011-10-10 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases
Keywords: PAD; CVA; ACS
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lifestyle counseling (Experimental): Group consultation and individual nurse consultation
  Interventions: Behavioral: Life style counseling; Behavioral: an individualized web portal; Behavioral: individual and group consultations
- e health (Experimental): An individual web based entry
  Interventions: Behavioral: an individualized web portal
- usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Life style counseling — A nurse-based intervention with face-to-face contacts based on motivational interviewing techniques and influence on behavioral determinants. Well-trained nurses in our hospital will apply these behavioral change interventions. An individual contact will take about twenty minutes.
  Arms: Lifestyle counseling
Behavioral: an individualized web portal — This website shows patient's lab results, life style issues, blood pressure and weight in various risk monitors. These lab results and lifestyle changes will be visualized in risk monitors and provide structural feedback to the patient. The results of the screening and the two additional visits can be seen by the patient.
  Arms: Lifestyle counseling; e health
Behavioral: individual and group consultations — group consultations with peers and a nurse individual consultation with a nurse
  Arms: Lifestyle counseling

SUMMARY:
The purpose of this study is to investigate whether a nurse-based intervention, consisting of structural informative consulting and motivational counseling, on top of usual care with or without personalized web-based visualization of cardiovascular risk levels, improves the medication adherence in high risk cardiovascular patients.

DETAILED DESCRIPTION:
Poor adherence to medication is one of the limitations in the treatment of cardiovascular disease. As a consequence the risk of premature death, hospital admissions and related costs is increasing. Therefore, detection of apparent poor adherence and interventions to improve adherence, are of great importance to enhance cardiovascular risk management over time.

This study is a prospective randomized trial, which compares 1) usual care with 2) the effect of a personalized visualization of cardiovascular risk levels (website) to support self management and 3) the additional effect of a communication intervention by a nurse on adherence on top of 2). Adherence is determined and continuously monitored with a dedicated calculation of refill data obtained from patient's pharmacy.

ELIGIBILITY:
Inclusion Criteria:

* All subsequent patients, included in the hospital-screening program with manifestations of atherosclerotic disease (acute coronary syndrome, peripheral arterial disease or stroke/TIA) or elevated cardiovascular risk due to hypertension, diabetes or hyperlipidemia.

Exclusion Criteria:

* Age below 18 years, actual pregnancy, problems with Dutch language or logistic problems, which may hinder intervention on adherence behavior. Severe co-morbidity, including mental handicap, according to their physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2011-11; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in degree of Adherence | Change from baseline in degree of Adherence at 12 month
  The degree of Adherence to medication for each group at 12 month from baseline, as calculated by prescription refill data

SECONDARY OUTCOMES:
Clinical outcome | Change from baseline in level of LDL-Cholesterol at 12 months
  Change in LDL-Cholesterol level in each group at 12 months from baseline
Clinical outcome | Change from baseline in Sytolic Blood Pressure at 12 months
  Change in Systolic Blood Pressure in each group at 12 months from baseline
Clinical outcome | Change from baseline in Body Mass Index at 12 months
  Change in Body Mass Index (BMI) in each group at 12 months from baseline
Clinical outcome | Change from baseline in Waist Circumference at 12 months
  Change in Waist Circumference in each group at 12 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bas JH Bredie, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University medical centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Sieben A, van Onzenoort HA, van Dulmen S, van Laarhoven C, Bredie SJ. A nurse-based intervention for improving medication adherence in cardiovascular patients: an evaluation of a randomized controlled trial. Patient Prefer Adherence. 2019 May 23;13:837-852. doi: 10.2147/PPA.S197481. eCollection 2019. PMID 31213778
- [Derived] Sieben A, van Onzenoort HA, van Laarhoven KJ, Bredie SJ. A Multifaceted Nurse- and Web-Based Intervention for Improving Adherence to Treatment in Patients With Cardiovascular Disease: Rationale and Design of the MIRROR Trial. JMIR Res Protoc. 2016 Sep 13;5(3):e187. doi: 10.2196/resprot.5750. PMID 27624877